CLINICAL TRIAL: NCT00156572
Title: Management of Hyponatremia in Preterm Infants on Diuretics
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: decreasing rate of enrollment
Sponsor: The University of Texas Health Science Center, Houston (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Hyponatremia-Diuretics
Record Dates: First submitted 2005-09-07; First posted 2005-09-12 (Estimated); Last update posted 2007-12-27 (Estimated); Status verified 2007-12

CONDITIONS: Bronchopulmonary Dysplasia; Hyponatremia on Diuretics
MeSH Terms: conditions — Bronchopulmonary Dysplasia

INTERVENTIONS:
Procedure: Sodium supplementation
Procedure: Fluid restriction

SUMMARY:
Hydrochlorothiazide and spironolactone are diuretics that are commonly in preterm infants with bronchopulmonary dysplasia (BPD). Hyponatremia (low blood salt) is a common side effect. It is uncertain whether the best way to treat the hyponatremia is by oral salt supplementation or restricting fluid intake. Our hypothesis is that fluid restricted infants will be better able to preserve the beneficial effects of diuretics on the lungs. The study will include very low birth weight infants (VLBW) 400-1500g from Hermann Memorial Children's Hospital NICU or LBJ General Hospital NICU with BPD. They will be enrolled and randomly assigned to either the salt supplementation group or the fluid restriction group once they become hyponatremic (defined as serum Na <130). The study intervention will take place for four weeks. The primary outcome will be assessed by comparing the patient's initial oxygen and breathing machine requirements with those at the end of the four-week study period.

DETAILED DESCRIPTION:
Study Question:

Among very low birth weight infants, 400-1500 g, with bronchopulmonary dysplasia who develop hyponatremia while receiving hydrochlorothiazide diuretics: does oral sodium supplementation compared to fluid restriction affect FiO2 requirements (change in Respiratory Index Score [RIS] in Ventilated or CPAP babies, or change in FiO2 in spontaneously breathing babies) after four weeks?

Randomization Method:

Enrolled patients will be randomly assigned to either the sodium supplementation group or the fluid restriction group once they become hyponatremic (serum sodium < 130) while taking hydrochlorothiazide.

Interventions:

Sodium Supplementation: Patients randomized to the sodium supplementation group will receive oral NaCl added to their feeds. When the serum sodium is 125-130, they will have 2 meq/kg/day of NaCl added to their feeds. If the serum sodium is 120-124, they will have 4 meq/kg/day of NaCl added to their feeds. Na supplementation will continue until the serum Na is >135.

Fluid Restriction: Patients randomized to the fluid restriction group will have fluid intake decreased by 20cc/kg/day. In order to maintain approximately the same caloric intake, 0.5 cc/kg/dose of corn oil (8.4kcal/cc), will be administered as a bolus every 6 hours. If this fluid restriction doesn't increase the serum sodium to above 130 within one week or if the serum Na is 120-124 and if the infant is receiving > 140 cc/kg/d, the fluid intake will be decreased by an additional 10cc/kg/day for one additional week.

Outcome Assessments Primary Outcome - the change in FiO2/RIS between baseline and outcome at 4 weeks after enrollment.

Secondary Outcomes

1. 24-hour urine sodium, calcium, and creatinine at 4 weeks.
2. The mean serum Na+ nadir for each group.
3. The mean serum K+ nadir for each group.
4. Time to extubation for infants ventilated at enrollment.
5. Time on CPAP or mechanical ventilation for infants on CPAP at enrollment.

Sample Size:

The estimated sample size for the study will be 58, based on an effect size of 10% if the mean FiO2 is 40% (0.1 x 40= 4% absolute difference), expected standard deviation of 5% for FiO2, alpha (two-sided) = 0.05; Beta = 1 - 0.80 = 0.20.

Analysis:

The following analysis plan has been designed to allow every randomized infant to be included in the analysis (intention-to-treat analysis) regardless of whether they are intubated, extubated, taken off or put onto CPAP, or if they die during the course of the 4-week study period. All infants (both study groups combined) will be assigned a rank at baseline and at outcome (4 weeks) within each of the following subgroups: infants on O2 by oxyhood, infants on nasal cannula, infants on CPAP, infants on the ventilator, infants who die during the study. For each infant, a change in rank (outcome minus baseline) will be calculated. The change in rank will be compared between the two study groups using a non-parametric test.

ELIGIBILITY:
Inclusion Criteria:

1. Very low birth weight infants, 400-1500 grams
2. Bronchopulmonary dysplasia defined by an oxygen requirement greater than 30% at 4 weeks of age and chest x-ray findings consistent with developing chronic lung disease.
3. Receiving 120kcal/kg/d enterally with fortified human milk or 24 kcal/oz formula
4. Hyponatremic (defined as serum Na <130).

Exclusion Criteria:

1. Known congenital anomalies involving the heart, lungs, kidneys, or chromosomal abnormalities.
2. Creatinine ≥ 1.3.
3. Enteral ostomy.

Ages: 4 Weeks to 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 58 (Estimated)
Dates: Start 2005-04; Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Oxygen and ventilator requirement expressed as RIS

SECONDARY OUTCOMES:
Urine sodium, calcium, creatinine, serum Na nadir, serum K nadir, duration of mechanical ventilation, duration of CPAP

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen A Kennedy, MD, MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- Memorial Hermann Children's Hospital, Houston, Texas, United States